CLINICAL TRIAL: NCT02805647
Title: Association Between Vitamin D Receptor Polymorphism and Serum Vitamin D Levels in Children With Low-Energy Fractures
Status: Completed | Type: Observational
Sponsor: Medical University of Bialystok (Other)
Collaborators: American Medical Holdings Inc., Staten Island, NY 10314 USA (Unknown); School of Pharmacy, Creighton University, Omaha, NE 68178 USA (Unknown)
Responsible Party: Principal Investigator, Michal Karpinski, MD, Medical University of Bialystok
Other Study IDs: MUBialystok
Record Dates: First submitted 2016-05-27; First posted 2016-06-20 (Estimated); Results first posted 2019-11-19 (Actual); Last update posted 2019-12-04 (Actual); Status verified 2019-11

CONDITIONS: Vitamin D Receptor Defect
Keywords: 25-Hydroxy-vitamin D, children, bone fractures, vitamin D receptor polymorphism
MeSH Terms: conditions — Fractures, Bone

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Fracture/study group: The study group consisted of 100 children aged 3 to 18 years (78% boys) hospitalized in the Department of Pediatric Orthopedics in 2011-2013 due to low-energy fractures
- Control group: The control group (122 children, 68% boys) consisted of children aged 3 to 17 years, hospitalized for other reasons (injuries, diagnosis of knee ligament injuries and others) without fractures

SUMMARY:
This study was designed to determine the impact of vitamin D serum levels and vitamin D receptor (VDR) polymorphisms on the occurrence of low energy fractures in children.

DETAILED DESCRIPTION:
The study group consisted of 100 children aged 3 to 18 years (78% boys) hospitalized in the Department of Pediatric Orthopedics in 2011-2013 due to low-energy fractures. The control group (122 children, 68% boys) consisted of children aged 3 to 17 years, hospitalized for other reasons (injuries, diagnosis of knee ligament injuries and others) without fractures. Children with osteogenesis imperfecta (OI) were excluded from the study. From each patient and their parent/guardian a written informed consent to participate in the study was obtained. Low-energy fracture was defined as a fracture sustained from a fall from the patient's own height or a fall during team games. All fractures were radiologically confirmed.

During hospitalization the patients and their parents completed a questionnaire on demographic data, the place of residence (urban/rural), earlier fractures and physical activity. The degree of sexual maturity was assessed using a survey of puberty development on the basis of Puberty Development Scale [20-22]. The patients' body weights and heights were measured, and the Cole indicator was calculated to assess the nutritional status of the patients.

Serum concentrations of total vitamin D [25-hydroxy vitamin D3 ((25(OH)D3)) plus 25-hydroxy vitamin D2 ((25(OH)D2))] in the plasma of all the children were determined by electrochemiluminescence using paramagnetic particles coated with streptavidin and ruthenium compound on the Cobas e 411 apparatus by Roche. According to our laboratory, the reference value range for total vitamin D was 30.0 - 74.0 ng/ml.Whole blood samples were collected in tubes containing EDTA and stored at -20°C. DNA was isolated using the MasterPureTM DNA Purification Kit (Akor Laboratories) and quantified on a spectrophotometer (Nanodrop 2000, Thermo Scientific). The genotypes for four restriction fragment length polymorphisms of the vitamin D receptor (VDR) gene were determined by standard polymerase chain reaction (PCR) techniques and enzymatic digestion of the products with FokI, ApaI, TaqI and BsmI (Thermo Scientific). In short, PCR were performed in a final volume of 20 µl containing 50-100 ng DNA, 0.3 µM of each primer and JumpStartTM REDTaqTM ReadyMixTM (Sigma). After initial denaturation for 3 min at 94 °C, samples were subjected to 35 cycles of amplification, consisting of a 30-sec denaturing phase at 94 °C, a 30-sec annealing phase (FokI at 60 °C, ApaI and TaqI at 70 °C, BsmI at 62 °C), a 30-s extension phase at 72 °C, and 4-min at 72 °C on a Bio-Rad thermal cycler CFX96TM. The primers used for FokI polymorphism were: forward 5'-AGC TGG CCC TGG CAC TGA CTC TGC TCT-3', reverse 5'-ATG GAA ACA CCT TGC TTC TTC TCC CTC-3'; ApaI and TaqI: forward 5'-CAG AGC ATG GAC AGG GAG CAA-3', reverse 5'-GCA ACT CCT CAT GGC TGA GGT CTC-3' and BsmI: forward 5'-AGT GTG CAG GCG ATT CGT AG-3', reverse 5'-ATA GGC AGA ACC ATC TCT CAG-3' [25]. The PCR products were digested according to the manufacturer's instructions and separated on 2% agarose gel. The polymorphisms were documented by photographing under UV illumination using G:Box (Syngene). A random subset (20% of samples) was repeated to verify the results. Upper case letters "F", "A", "T" and "B" indicate the absence of the cut site for FokI, ApaI, TaqI and BsmI polymorphisms, respectively, whereas lower case letters "f", "a", "t", and "b" indicate its presence.To examine the relationships between quality attributes Chi-square test of independence and Fisher's exact test were used. The normality of distribution was verified using the Kolmogorov-Smirnov test with the Lilliefors significance correction and the Shapiro-Wilk test. There was no normal distribution of quantitative variables analyzed. To compare the quantitative variables without normal distribution a nonparametric Mann - Whitney U test was used. Models of uni-variate and multi-variate linear regression and logistic regression were established. Results were considered statistically significant at p <0.05. The calculations were performed using Statistica 10.0 by StatSoft, IBM SPSS Statistics 21.0 by Predictive Solutions Company and Stata / IC 13.1 packages by StataCorp LP

ELIGIBILITY:
Inclusion Criteria:

* low-energy fractures.
* healthy children hospitalized for other reasons than fractures (injuries, diagnosis of knee ligament injuries and others) without fractures

Exclusion Criteria:

* Children with osteogenesis imperfecta (OI) were excluded from the study.

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Study Group: Healthy children with low energy fractures Control group: Healthy children without fractures
Sampling Method: Probability Sample
Enrollment: 222 (Actual)
Dates: Start 2011-01; Primary Completion 2013-12 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michał Karpiński, MD, Principal Investigator — Department of Pediatric Orthopedics and Traumatology Medical University of Bialystok
Locations (1):
- Department of Pediatric Orthopedics and Traumatology Medical University of Bialystok, Bialystok, Poland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Jones IE, Williams SM, Dow N, Goulding A. How many children remain fracture-free during growth? a longitudinal study of children and adolescents participating in the Dunedin Multidisciplinary Health and Development Study. Osteoporos Int. 2002 Dec;13(12):990-5. doi: 10.1007/s001980200137. PMID 12459942
- [Background] Ma D, Jones G. Soft drink and milk consumption, physical activity, bone mass, and upper limb fractures in children: a population-based case-control study. Calcif Tissue Int. 2004 Oct;75(4):286-91. doi: 10.1007/s00223-004-0274-y. Epub 2004 Jul 30. PMID 15549642
- [Background] Wyshak G, Frisch RE. Carbonated beverages, dietary calcium, the dietary calcium/phosphorus ratio, and bone fractures in girls and boys. J Adolesc Health. 1994 May;15(3):210-5. doi: 10.1016/1054-139x(94)90506-1. PMID 8075091
- [Background] Carey DE, Golden NH. Bone Health in Adolescence. Adolesc Med State Art Rev. 2015 Aug;26(2):291-325. PMID 26999874
- [Background] Manning Ryan L, Teach SJ, Searcy K, Singer SA, Wood R, Wright JL, Hunting KL, Chamberlain JM. The Association Between Weight Status and Pediatric Forearm Fractures Resulting From Ground-Level Falls. Pediatr Emerg Care. 2015 Dec;31(12):835-8. doi: 10.1097/PEC.0000000000000628. PMID 26583933
- [Background] Yao Y, Zhu L, He L, Duan Y, Liang W, Nie Z, Jin Y, Wu X, Fang Y. A meta-analysis of the relationship between vitamin D deficiency and obesity. Int J Clin Exp Med. 2015 Sep 15;8(9):14977-84. eCollection 2015. PMID 26628980
- [Background] Thompson RM, Dean DM, Goldberg S, Kwasny MJ, Langman CB, Janicki JA. Vitamin D Insufficiency and Fracture Risk in Urban Children. J Pediatr Orthop. 2017 Sep;37(6):368-373. doi: 10.1097/BPO.0000000000000697. PMID 26600296
- [Background] Huber AM, Ward LM. The impact of underlying disease on fracture risk and bone mineral density in children with rheumatic disorders: A review of current literature. Semin Arthritis Rheum. 2016 Aug;46(1):49-63. doi: 10.1016/j.semarthrit.2016.02.003. Epub 2016 Feb 26. PMID 27020068
- [Background] Mohammadi Z, Fayyazbakhsh F, Ebrahimi M, Amoli MM, Khashayar P, Dini M, Zadeh RN, Keshtkar A, Barikani HR. Association between vitamin D receptor gene polymorphisms (Fok1 and Bsm1) and osteoporosis: a systematic review. J Diabetes Metab Disord. 2014 Oct 17;13(1):98. doi: 10.1186/s40200-014-0098-x. eCollection 2014. PMID 25364703
- [Background] Haussler MR, Whitfield GK, Haussler CA, Hsieh JC, Thompson PD, Selznick SH, Dominguez CE, Jurutka PW. The nuclear vitamin D receptor: biological and molecular regulatory properties revealed. J Bone Miner Res. 1998 Mar;13(3):325-49. doi: 10.1359/jbmr.1998.13.3.325. No abstract available. PMID 9525333
- [Background] Deluca HF, Cantorna MT. Vitamin D: its role and uses in immunology. FASEB J. 2001 Dec;15(14):2579-85. doi: 10.1096/fj.01-0433rev. PMID 11726533
- [Background] Szymczak I, Pawliczak R. The Active Metabolite of Vitamin D3 as a Potential Immunomodulator. Scand J Immunol. 2016 Feb;83(2):83-91. doi: 10.1111/sji.12403. PMID 26678915
- [Background] Hii CS, Ferrante A. The Non-Genomic Actions of Vitamin D. Nutrients. 2016 Mar 2;8(3):135. doi: 10.3390/nu8030135. PMID 26950144
- [Background] Holick MF. High prevalence of vitamin D inadequacy and implications for health. Mayo Clin Proc. 2006 Mar;81(3):353-73. doi: 10.4065/81.3.353. PMID 16529140
- [Background] Holick MF, Chen TC. Vitamin D deficiency: a worldwide problem with health consequences. Am J Clin Nutr. 2008 Apr;87(4):1080S-6S. doi: 10.1093/ajcn/87.4.1080S. PMID 18400738
- [Background] Ryan LM, Brandoli C, Freishtat RJ, Wright JL, Tosi L, Chamberlain JM. Prevalence of vitamin D insufficiency in African American children with forearm fractures: a preliminary study. J Pediatr Orthop. 2010 Mar;30(2):106-9. doi: 10.1097/BPO.0b013e3181d076a3. PMID 20179554
- [Background] Karpiński M, Popko J, Żelazowska-Rutkowska B.Prevalence of vitamin D insufficiency in children with low-energy fractures. Endokrynol Ped 2:9-16, 2011.
- [Background] Schilling S, Wood JN, Levine MA, Langdon D, Christian CW. Vitamin D status in abused and nonabused children younger than 2 years old with fractures. Pediatrics. 2011 May;127(5):835-41. doi: 10.1542/peds.2010-0533. Epub 2011 Apr 11. PMID 21482609
- [Background] Bond L, Clements J, Bertalli N, Evans-Whipp T, McMorris BJ, Patton GC, Toumbourou JW, Catalano RF. A comparison of self-reported puberty using the Pubertal Development Scale and the Sexual Maturation Scale in a school-based epidemiologic survey. J Adolesc. 2006 Oct;29(5):709-20. doi: 10.1016/j.adolescence.2005.10.001. Epub 2005 Dec 1. PMID 16324738
- [Background] Carskadon MA, Acebo C. A self-administered rating scale for pubertal development. J Adolesc Health. 1993 May;14(3):190-5. doi: 10.1016/1054-139x(93)90004-9. PMID 8323929
- [Background] Dick MD, Rose JR, Pulkkinen L, . Kaprio J. Measuring puberty and understanding its impact: A longitudinal study of adolescent twins. J Youth Adolesc 30:385-399, 2001.
- [Background] Cole TJ, Bellizzi MC, Flegal KM, Dietz WH. Establishing a standard definition for child overweight and obesity worldwide: international survey. BMJ. 2000 May 6;320(7244):1240-3. doi: 10.1136/bmj.320.7244.1240. PMID 10797032
- [Background] Cole TJ. The evidential value of developmental age imaging for assessing age of majority. Ann Hum Biol. 2015;42(4):379-88. doi: 10.3109/03014460.2015.1031826. Epub 2015 Jul 2. PMID 26133364
- [Background] Gyorffy B, Vasarhelyi B, Krikovszky D, Madacsy L, Tordai A, Tulassay T, Szabo A. Gender-specific association of vitamin D receptor polymorphism combinations with type 1 diabetes mellitus. Eur J Endocrinol. 2002 Dec;147(6):803-8. doi: 10.1530/eje.0.1470803. PMID 12457456
- [Background] Marshall WA, Tanner JM. Variations in pattern of pubertal changes in girls. Arch Dis Child. 1969 Jun;44(235):291-303. doi: 10.1136/adc.44.235.291. No abstract available. PMID 5785179
- [Background] Marshall WA, Tanner JM. Variations in the pattern of pubertal changes in boys. Arch Dis Child. 1970 Feb;45(239):13-23. doi: 10.1136/adc.45.239.13. PMID 5440182
- [Background] Lyons RA, Sellstrom E, Delahunty AM, Loeb M, Varilo S. Incidence and cause of fractures in European districts. Arch Dis Child. 2000 Jun;82(6):452-5. doi: 10.1136/adc.82.6.452. PMID 10833175
- [Background] Hansson G, Hirsch G. Fractures in children. J Pediatr Orthop B. 1997 Apr;6(2):77-8. doi: 10.1097/01202412-199704000-00001. No abstract available. PMID 9165434
- [Background] Goulding A, Jones IE, Taylor RW, Manning PJ, Williams SM. More broken bones: a 4-year double cohort study of young girls with and without distal forearm fractures. J Bone Miner Res. 2000 Oct;15(10):2011-8. doi: 10.1359/jbmr.2000.15.10.2011. PMID 11028455
- [Background] Goulding A, Grant AM, Williams SM. Bone and body composition of children and adolescents with repeated forearm fractures. J Bone Miner Res. 2005 Dec;20(12):2090-6. doi: 10.1359/JBMR.050820. Epub 2005 Aug 22. PMID 16294262
- [Background] Goulding A, Rockell JE, Black RE, Grant AM, Jones IE, Williams SM. Children who avoid drinking cow's milk are at increased risk for prepubertal bone fractures. J Am Diet Assoc. 2004 Feb;104(2):250-3. doi: 10.1016/j.jada.2003.11.008. PMID 14760576
- [Background] Clark EM, Tobias JH, Ness AR. Association between bone density and fractures in children: a systematic review and meta-analysis. Pediatrics. 2006 Feb;117(2):e291-7. doi: 10.1542/peds.2005-1404. PMID 16452336
- [Background] Ferrari SL, Chevalley T, Bonjour JP, Rizzoli R. Childhood fractures are associated with decreased bone mass gain during puberty: an early marker of persistent bone fragility? J Bone Miner Res. 2006 Apr;21(4):501-7. doi: 10.1359/jbmr.051215. Epub 2006 Apr 5. PMID 16598368
- [Background] Abrams SA, Griffin IJ, Hawthorne KM, Chen Z, Gunn SK, Wilde M, Darlington G, Shypailo RJ, Ellis KJ. Vitamin D receptor Fok1 polymorphisms affect calcium absorption, kinetics, and bone mineralization rates during puberty. J Bone Miner Res. 2005 Jun;20(6):945-53. doi: 10.1359/JBMR.050114. Epub 2005 Jan 31. PMID 15883634
- [Background] Macdonald HM, McGuigan FE, Stewart A, Black AJ, Fraser WD, Ralston S, Reid DM. Large-scale population-based study shows no evidence of association between common polymorphism of the VDR gene and BMD in British women. J Bone Miner Res. 2006 Jan;21(1):151-62. doi: 10.1359/JBMR.050906. Epub 2005 Sep 12. PMID 16355284
- [Background] Ji GR, Yao M, Sun CY, Li ZH, Han Z. BsmI, TaqI, ApaI and FokI polymorphisms in the vitamin D receptor (VDR) gene and risk of fracture in Caucasians: a meta-analysis. Bone. 2010 Sep;47(3):681-6. doi: 10.1016/j.bone.2010.06.024. Epub 2010 Jun 28. PMID 20601302
- [Background] Uitterlinden AG, Ralston SH, Brandi ML, Carey AH, Grinberg D, Langdahl BL, Lips P, Lorenc R, Obermayer-Pietsch B, Reeve J, Reid DM, Amedei A, Bassiti A, Bustamante M, Husted LB, Diez-Perez A, Dobnig H, Dunning AM, Enjuanes A, Fahrleitner-Pammer A, Fang Y, Karczmarewicz E, Kruk M, van Leeuwen JP, Mavilia C, van Meurs JB, Mangion J, McGuigan FE, Pols HA, Renner W, Rivadeneira F, van Schoor NM, Scollen S, Sherlock RE, Ioannidis JP; APOSS Investigators; EPOS Investigators; EPOLOS Investigators; FAMOS Investigators; LASA Investigators; Rotterdam Study Investigators; GENOMOS Study. The association between common vitamin D receptor gene variations and osteoporosis: a participant-level meta-analysis. Ann Intern Med. 2006 Aug 15;145(4):255-64. doi: 10.7326/0003-4819-145-4-200608150-00005. PMID 16908916
- [Background] Uitterlinden AG, Fang Y, Van Meurs JB, Pols HA, Van Leeuwen JP. Genetics and biology of vitamin D receptor polymorphisms. Gene. 2004 Sep 1;338(2):143-56. doi: 10.1016/j.gene.2004.05.014. PMID 15315818
- [Background] Fang Y, Rivadeneira F, van Meurs JB, Pols HA, Ioannidis JP, Uitterlinden AG. Vitamin D receptor gene BsmI and TaqI polymorphisms and fracture risk: a meta-analysis. Bone. 2006 Oct;39(4):938-45. doi: 10.1016/j.bone.2006.04.016. PMID 16769262
- [Background] Horst-Sikorska W, Kalak R, Wawrzyniak A, Marcinkowska M, Celczynska-Bajew L, Slomski R. Association analysis of the polymorphisms of the VDR gene with bone mineral density and the occurrence of fractures. J Bone Miner Metab. 2007;25(5):310-9. doi: 10.1007/s00774-007-0769-5. Epub 2007 Aug 25. PMID 17704996
- [Background] Bener A, Al-Ali M, Hoffmann GF. Vitamin D deficiency in healthy children in a sunny country: associated factors. Int J Food Sci Nutr. 2009;60 Suppl 5:60-70. doi: 10.1080/09637480802400487. Epub 2008 Oct 22. PMID 18946796
- [Background] Steele B, Serota A, Helfet DL, Peterson M, Lyman S, Lane JM. Vitamin D deficiency: a common occurrence in both high-and low-energy fractures. HSS J. 2008 Sep;4(2):143-8. doi: 10.1007/s11420-008-9083-6. Epub 2008 Jul 19. PMID 18815858
- [Background] Peters BS, dos Santos LC, Fisberg M, Wood RJ, Martini LA. Prevalence of vitamin D insufficiency in Brazilian adolescents. Ann Nutr Metab. 2009;54(1):15-21. doi: 10.1159/000199454. Epub 2009 Feb 5. PMID 19194104
- [Background] Turner AG, Anderson PH, Morris HA. Vitamin D and bone health. Scand J Clin Lab Invest Suppl. 2012;243:65-72. doi: 10.3109/00365513.2012.681963. PMID 22536765
- [Background] Becker C, Crow S, Toman J, Lipton C, McMahon DJ, Macaulay W, Siris E. Characteristics of elderly patients admitted to an urban tertiary care hospital with osteoporotic fractures: correlations with risk factors, fracture type, gender and ethnicity. Osteoporos Int. 2006;17(3):410-6. doi: 10.1007/s00198-005-0001-1. Epub 2005 Nov 8. PMID 16283067
- [Background] Glowacki J, Hurwitz S, Thornhill TS, Kelly M, LeBoff MS. Osteoporosis and vitamin-D deficiency among postmenopausal women with osteoarthritis undergoing total hip arthroplasty. J Bone Joint Surg Am. 2003 Dec;85(12):2371-7. doi: 10.2106/00004623-200312000-00015. PMID 14668507
- [Background] Janssen HC, Samson MM, Verhaar HJ. Vitamin D deficiency, muscle function, and falls in elderly people. Am J Clin Nutr. 2002 Apr;75(4):611-5. doi: 10.1093/ajcn/75.4.611. PMID 11916748
- [Background] Hitz MF, Jensen JE, Eskildsen PC. Bone mineral density and bone markers in patients with a recent low-energy fracture: effect of 1 y of treatment with calcium and vitamin D. Am J Clin Nutr. 2007 Jul;86(1):251-9. doi: 10.1093/ajcn/86.1.251. PMID 17616788
- [Background] Pawley N, Bishop NJ. Prenatal and infant predictors of bone health: the influence of vitamin D. Am J Clin Nutr. 2004 Dec;80(6 Suppl):1748S-51S. doi: 10.1093/ajcn/80.6.1748S. PMID 15585799
- [Background] Lehtonen-Veromaa MK, Mottonen TT, Nuotio IO, Irjala KM, Leino AE, Viikari JS. Vitamin D and attainment of peak bone mass among peripubertal Finnish girls: a 3-y prospective study. Am J Clin Nutr. 2002 Dec;76(6):1446-53. doi: 10.1093/ajcn/76.6.1446. PMID 12450915
- [Background] Li K, Shi Q, Yang L, Li X, Liu L, Wang L, Li Q, Wang G, Li CY, Gao TW. The association of vitamin D receptor gene polymorphisms and serum 25-hydroxyvitamin D levels with generalized vitiligo. Br J Dermatol. 2012 Oct;167(4):815-21. doi: 10.1111/j.1365-2133.2012.11132.x. PMID 22762534
- [Background] Santos BR, Mascarenhas LP, Satler F, Boguszewski MC, Spritzer PM. Vitamin D deficiency in girls from South Brazil: a cross-sectional study on prevalence and association with vitamin D receptor gene variants. BMC Pediatr. 2012 Jun 8;12:62. doi: 10.1186/1471-2431-12-62. PMID 22681928
- [Background] Clark EM, Ness AR, Tobias JH. Vigorous physical activity increases fracture risk in children irrespective of bone mass: a prospective study of the independent risk factors for fractures in healthy children. J Bone Miner Res. 2008 Jul;23(7):1012-22. doi: 10.1359/jbmr.080303. PMID 18570539
- [Background] Manias K, McCabe D, Bishop N. Fractures and recurrent fractures in children; varying effects of environmental factors as well as bone size and mass. Bone. 2006 Sep;39(3):652-7. doi: 10.1016/j.bone.2006.03.018. Epub 2006 Jun 12. PMID 16765659
- [Result] Landin LA. Fracture patterns in children. Analysis of 8,682 fractures with special reference to incidence, etiology and secular changes in a Swedish urban population 1950-1979. Acta Orthop Scand Suppl. 1983;202:1-109. PMID 6574687

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Children with low energy fractures
Pre-assignment Details: without bone diseases such as OI
Period: Overall Study
Arm/Group | Fracture/Study Group | Control Group
Started | 100 (at the moment of submision) | 122 (at the moment of submision)
Completed | 100 (after laboratory tests) | 122 (after laboratory tests)
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Children with low energy fractures without bone diseases in study group and children without history of fractures in control group
Groups:
- Total: Total of all reporting groups
Arm/Group | Fracture/Study Group | Control Group | Total
Number analyzed (Participants) | 100 | 122 | 222
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 100 | 122 | 222
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Standard Deviation); unit: years] | 13 (2) | 13 (2) | 13 (2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 39 | 61
  Male | 78 | 83 | 161
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants] — Polish Children of Podlasie region
  participants
    Poland | 100 | 122 | 222
Total vitamin D [25(OH)D3 plus 25(OH)D2] serum concentrations were evaluated in every patient. Genot [Median (Standard Deviation); unit: ng/ml] | 13.81 (12) | 17.49 (16) | 15 (14)

OUTCOME MEASURES:

1. Primary Outcome: Vitamin D Status; VDR Status
Description: Serum concentrations of total vitamin D; VDR polymorphism test
Time Frame: We measured Vitamin D status at the time of admission - at the time of fracture
Population: Children from Poland Podlasie region
Measure: Mean (Inter-Quartile Range); unit: ng/ml
Arm/Group | Fracture/Study Group | Control Group
Number analyzed (Participants) | 100 | 122
ng/ml | 13.81 [8 to 18] | 17.49 [11 to 23]

ADVERSE EVENTS:
Time Frame: We measured vitamin D status and VDR polymporphism at admission to hospital and when patients were enrolled to the study
Arm/Group | Fracture/Study Group | Control Group
Serious Adverse Events (participants affected / at risk) | 0/100 | 0/122
Other Adverse Events (participants affected / at risk) | 0/100 | 0/122

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No